CLINICAL TRIAL: NCT04993677
Title: An Open-label, Phase 2 Basket Study of SEA-CD40 Combination Therapies in Advanced Malignancies
Brief Title: A Study of SEA-CD40 Given With Other Drugs in Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNS40-002; KEYNOTE-C86 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Melanoma; Carcinoma, Non-Small- Cell Lung
Keywords: Relapsed melanoma; Refractory melanoma; Metastatic uveal melanoma; Metastatic PD-(L)1-naïve melanoma; Non-squamous NSCLC; NSCLC; Non-small cell lung cancer; Seattle Genetics
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Uveal Melanoma | interventions — pembrolizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melanoma Arm (Experimental): SEA-CD40 + pembrolizumab
  Interventions: Drug: SEA-CD40; Drug: pembrolizumab (KEYTRUDA®)
- NSCLC Arm (Experimental): SEA-CD40 + pembrolizumab + pemetrexed + carboplatin
  Interventions: Drug: SEA-CD40; Drug: pembrolizumab (KEYTRUDA®); Drug: pemetrexed; Drug: carboplatin

INTERVENTIONS:
Drug: SEA-CD40 — Given into the vein (IV; intravenously); schedule is cohort-specific
Drug: pembrolizumab (KEYTRUDA®) — Given by IV; schedule is cohort-specific.
Drug: pemetrexed — Given by IV on Day 1 of each 21-day cycle.
  Other Names: Alimta
  Arms: NSCLC Arm
Drug: carboplatin — Given by IV on Day 1 of Cycles 1-4. Each cycle will be 21 days long.
  Other Names: Paraplatin
  Arms: NSCLC Arm

SUMMARY:
This trial is being done to see if an experimental drug (SEA-CD40) works when it's given with other cancer drugs to treat some types of cancer. It will also study side effects from the drug.

There are 2 parts in this trial. In one part, participants have melanoma that has come back after treatment or can't be removed by surgery. Participants in this part will get SEA-CD40 and pembrolizumab. In the other part, participants have non-small cell lung cancer (NSCLC) that has spread through their body. These participants will get SEA-CD40, pembrolizumab, carboplatin, and pemetrexed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable malignancy defined as one of the following:

  * Cohort 1: Relapsed and/or refractory metastatic melanoma

    * Uveal/ocular melanoma is excluded
    * Must have progressed on treatment with an anti-PD-(L)1 mAb. PD-(L)1 treatment progression is defined as meeting all of the following criteria:

      * Has received at least 2 doses of an approved anti-PD-(L)1 mAb
      * Has demonstrated disease progression after PD-(L)1 as defined by RECIST v1.1.
      * Progressive disease has been documented within 12 weeks from the last dose of anti- PD-(L)1 mAb
      * Last dose of anti-PD-(L)1 must have been within 90 days prior to enrollment
    * Participants with a targetable BRAF mutation must have been treated with, been intolerant of, or declined treatment with BRAF/MEK targeted therapy prior to study entry
  * Cohort 2: Metastatic uveal melanoma

    * Must not have received prior treatment for advanced or metastatic disease except for prior adjuvant/neoadjuvant immunotherapy
    * No prior liver-directed therapy
  * Cohort 3: Metastatic PD-(L)1-naive melanoma

    * Uveal/ocular melanoma is excluded
    * Must not have received prior treatment for advanced or metastatic disease except for prior adjuvant/neoadjuvant immunotherapy.
    * For participants with a targetable BRAF mutation, prior BRAF/MEK targeted therapy is allowed if completed 4 weeks prior to first dose of study treatment.
  * Cohorts 4 and 5: Non-squamous NSCLC

    * Participants must have stage IV disease per AJCC 8th edition
    * No known driver mutations/alterations mutation for which targeted therapy is available
    * Must have non-squamous histology.
    * No prior therapy for metastatic disease
    * No prior treatment with anti-PD-(L)1 or PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms
* Able to provide archival tumor tissue from locations not radiated prior to biopsy. If archival tumor sample is not available a fresh baseline biopsy is required.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Measurable disease per RECIST v1.1 at baseline

Exclusion Criteria:

* History of another malignancy within 3 years of first dose of study drug
* Active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Previous exposure to CD40-targeted therapy
* Currently on chronic systemic steroids in excess of physiologic replacement
* Has had an allogeneic tissue/solid organ transplant.
* History of autoimmune disease that has required systemic treatment in the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hayman, MD, Study Director — Seagen Inc.
Locations (29):
- United States (23):
  - Highlands Oncology Group, Springdale, Arkansas
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - California Pacific Medical Center Research Institute/Sutter Medical Centre, San Francisco, California
  - University of California at San Francisco, San Francisco, California
  - Florida Cancer Specialists - South Region, Fort Myers, Florida
  - Florida Cancer Specialists - North Region, St. Petersburg, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Community Health Network, Indianapolis, Indiana
  - American Oncology Networks LLC, Baton Rouge, Louisiana
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Regions Cancer Care Center, Saint Paul, Minnesota
  - Morristown Medical Center/ Carol G. Simon Cancer Center, Morristown, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center Research, LLC, Canton, Ohio
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Kaiser Permanente Oregon, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Tennessee Oncology-Nashville/Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern/Simmons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Carbone Cancer Center / University of Wisconsin, Madison, Wisconsin
- CHU de Quebec-Universite Laval, Québec, Canada
- Hopital Foch, Suresnes, Other, France
- Universitatsklinikum Heidelberg, Heidelberg, Other, Germany
- Spain (2):
  - START Madrid-CIOCC_Hospital HM Sanchinarro, Madrid, Other
  - Hospital Clinico Universitario de Valencia, Valencia, Other
- Karolinska University Hospital, Stockholm, Other, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study planned to have 5 cohorts-Cohort 1: relapsed/refractory melanoma, Cohort 2: uveal melanoma, Cohort 3: programmed cell death 1 ligand 1 (PD-[L]1)-naive melanoma, Cohort 4: non-small cell lung cancer (NSCLC), programmed cell death ligand 1 (PD-L1) 1-49%, Cohort 5: NSCLC, PD-L1 < 1%. No participant was enrolled and treated in Cohort 3.
Pre-assignment Details: "Study termination by sponsor" was used as end of study reason as long-term follow-up was discontinued following decision to close enrollment. Study status is listed completed as participants were permitted to receive treatment until they met protocol defined reasons to stop. After treatment discontinuation, participants were followed through duration of safety reporting period, and then ended study as no further disease or survival follow-up was required.
Groups:
- Cohort 1: Relapsed/Refractory Melanoma: Participants with relapsed/refractory melanoma, were administered SEA-CD40 10 micrograms per kilogram (mcg/kg) as an intravenous (IV) infusion on Day 1 and Day 22 of 42-day cycles along with Pembrolizumab 400 milligrams (mg) as an IV infusion on Day 8 of 42-day cycles.
- Cohort 2: Uveal Melanoma: Participants with uveal melanoma, were administered SEA-CD40 10 mcg/kg as an IV infusion on Day 1 and Day 22 of 42-day cycles along with Pembrolizumab 400 mg as an IV infusion on Day 8 of 42-day cycles.
- Cohort 4: NSCLC, PD-L1 1-49%: Participants with NSCLC, PD-L1 1-49%, were administered SEA-CD40 10 mcg/kg as an IV infusion on Day 3 of 21-day cycles along with Pembrolizumab 200 mg as an IV infusion on Day 1 of 21-day cycles and Pemetrexed 500 mg per meter square (/m^2) as an IV infusion on Day 1 of 21-day cycles and Carboplatin area under curve (AUC) 5 milligrams/milliliter/minute (mg/mL/min) as an IV infusion on Day 1 of 21-day (Cycles 1-4).
- Cohort 5: NSCLC, PD-L1 < 1%: Participants with NSCLC, PD-L1 <1%, were administered SEA-CD40 10 mcg/kg as an IV infusion on Day 3 of 21-day cycles along with Pembrolizumab 200 mg as an IV infusion on Day 1 of 21-day cycles and Pemetrexed 500 mg/m^2 as an IV infusion on Day 1 of 21-day cycles and Carboplatin AUC 5 mg/mL/min as an IV infusion on Day 1 of 21-day (Cycles 1-4).
Period: Overall Study
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Started | 21 | 39 | 9 | 8
Completed | 0 | 0 | 0 | 0
Not Completed | 21 | 39 | 9 | 8
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Death | 11 | 8 | 3 | 1
Not completed — Subject withdrawal of consent | 4 | 3 | 0 | 2
Not completed — Study termination by sponsor | 3 | 25 | 3 | 3
Not completed — Other | 2 | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received any amount of study drug.
Groups:
- Cohort 1: Relapsed/Refractory Melanoma: Participants with relapsed/refractory melanoma, were administered SEA-CD40 10 mcg/kg as an IV infusion on Day 1 and Day 22 of 42-day cycles along with Pembrolizumab 400 mg as an IV infusion on Day 8 of 42-day cycles.
- Cohort 4: NSCLC, PD-L1 1-49%: Participants with NSCLC, PD-L1 1-49%, were administered SEA-CD40 10 mcg/kg as an IV infusion on Day 3 of 21-day cycles along with Pembrolizumab 200 mg as an IV infusion on Day 1 of 21-day cycles and Pemetrexed 500 mg/m^2 as an IV infusion on Day 1 of 21-day cycles and Carboplatin AUC 5 mg/mL/min as an IV infusion on Day 1 of 21-day (Cycles 1-4).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1% | Total
Number analyzed (Participants) | 21 | 39 | 9 | 8 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (11.6) | 62.3 (12.4) | 64.6 (9.2) | 66.8 (9.5) | 63.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 20 | 4 | 2 | 35
  Male | 12 | 19 | 5 | 6 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 1 | 4
  Not Hispanic or Latino | 16 | 38 | 9 | 5 | 68
  Unknown or Not Reported | 2 | 1 | 0 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 16 | 39 | 9 | 5 | 69
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 0 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (cORR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Per Investigator Assessment
Description: cORR is defined as the percentage of participants achieving a confirmed complete response (CR) or partial response (PR) according to RECIST v1.1. CR: disappearance of all target, non-target lesions, all lymph nodes must be non-pathological in size (<10 millimeter [mm] short axis), PR: at least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters persistence of one or more non-target lesions.
Time Frame: From start of study treatment until CR or PR (maximum up to 15.2 months)
Population: The response evaluable (RE) analysis set included all participants with measurable disease at baseline who received any amount of study drug and had at least one post-baseline disease assessment per RECIST v1.1 or discontinued study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Number analyzed (Participants) | 21 | 39 | 9 | 8
Percentage of participants | 0 [NA to NA] — The upper and lower limit of 95% CI was not estimable since no participant had event. | 5 [0.6 to 17.3] | 44 [13.7 to 78.8] | 25 [3.2 to 65.1]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Related TEAEs, Greater Than or Equal to (>=) Grade 3 TEAEs, Treatment Emergent Serious Adverse Event (TESAE), Treatment Related TESAE
Description: Adverse event (AE):untoward medical occurrence in participant/clinical investigational participant administered medicinal product which doesn't necessarily have causal relationship with treatment. Serious AE (SAE):any AE that at any dose resulted in death, life threatening, required hospitalization/prolongation of hospitalization, disabling/incapacitating, congenital anomaly/birth defects.AEs included SAEs,non-SAEs.TEAEs:newly occurring/worsening after 1st dose of treatment.Treatment related TEAEs:related to treatment;relatedness judged by investigator. TEAEs graded according to National Cancer Institute Common Terminology Criteria for AEs (NCI-CTCAE) v4.03 (grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threating, grade 5=fatal). TESAEs:any TEAE that at any dose suspected to cause death, life-threatening, required hospitalization, disabling/incapacitating, congenital anomaly/birth defect. Treatment related TESAEs:related to treatment; relatedness judged by investigator.
Time Frame: From first dose of the study treatment (Day 1) up to approximately 18.5 months
Population: The safety analysis set included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Number analyzed (Participants) | 21 | 39 | 9 | 8
Participants
  TEAE | 17 | 37 | 8 | 8
  Treatment-related TEAE | 16 | 32 | 8 | 8
  >= Grade 3 TEAEs | 7 | 7 | 7 | 6
  TESAE | 4 | 5 | 5 | 5
  Treatment-related TESAE | 2 | 2 | 3 | 3

3. Secondary Outcome: Number of Participants With Grade Shift From Baseline to Maximum Post-Baseline in Serum Chemistry Laboratory Abnormalities Assessed by NCI CTCAE
Description: In this outcome measure, number of participants with baseline laboratory chemistry values as per NCI-CTCAE grade (grade 0=within normal limits, grade 1=mild, grade 2=moderate, grade 3=severe, grade 4= life-threatening) and corresponding changes or shift to the worst CTC grades post baseline were presented. Laboratory parameters evaluated: alanine aminotransferase increased, albumin decreased, alkaline phosphatase increased, aspartate aminotransferase increased, calcium corrected for albumin, creatinine increased, glomerular filtration rate (GFR) estimated decreased, glucose decreased, lactate dehydrogenase increased, potassium, sodium, total bilirubin increased. Baseline was defined as last non-missing grade before first dose of study treatment and worst post-baseline value defined as worst value post study treatment. Only those categories in which at least 1 participant had data in any reporting group were reported.
Time Frame: Baseline up to approximately 15.8 months
Population: The safety analysis set included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Number analyzed (Participants) | 21 | 39 | 9 | 8
Participants
  Alanine aminotransferase - increased: baseline Grade 0 to maximum post-baseline Grade 1 | 2 | 7 | 3 | 3
  Alanine aminotransferase - increased: baseline Grade 0 to maximum post-baseline Grade 2 | 0 | 3 | 1 | 0
  Alanine aminotransferase - increased: baseline Grade 0 to maximum post-baseline Grade 3 | 0 | 1 | 0 | 0
  Alanine aminotransferase - increased: baseline Grade 1 to maximum post-baseline Grade 0 | 0 | 1 | 0 | 0
  Alanine aminotransferase - increased: baseline Grade 2 to maximum post-baseline Grade 0 | 0 | 1 | 0 | 0
  Albumin - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 5 | 2 | 2 | 1
  Albumin - decreased: baseline Grade 0 to maximum post-baseline Grade 2 | 1 | 0 | 1 | 1
  Albumin - decreased: baseline Grade 1 to maximum post-baseline Grade 2 | 3 | 1 | 1 | 1
  Alkaline phosphatase - increased: baseline Grade 0 to maximum post-baseline Grade 1 | 4 | 9 | 1 | 1
  Alkaline phosphatase - increased: baseline Grade 1 to maximum post-baseline Grade 0 | 1 | 3 | 1 | 2
  Alkaline phosphatase - increased: baseline Grade 1 to maximum post-baseline Grade 2 | 1 | 0 | 0 | 0
  Alkaline phosphatase - increased: baseline Grade 2 to maximum post-baseline Grade 0 | 0 | 0 | 1 | 0
  Aspartate aminotransferase - increased: baseline Grade 0 to maximum post-baseline Grade 1 | 5 | 14 | 3 | 4
  Aspartate aminotransferase - increased: baseline Grade 0 to maximum post-baseline Grade 2 | 1 | 2 | 1 | 0
  Aspartate aminotransferase - increased: baseline Grade 1 to maximum post-baseline Grade 0 | 0 | 2 | 0 | 0
  Aspartate aminotransferase - increased: baseline Grade 1 to maximum post-baseline Grade 2 | 0 | 1 | 0 | 0
  Calcium corrected for albumin - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 2 | 1 | 4 | 1
  Calcium corrected for albumin - decreased: baseline Grade 0 to maximum post-baseline Grade 2 | 0 | 0 | 1 | 2
  Calcium corrected for albumin - decreased: baseline Grade 2 to maximum post-baseline Grade 1 | 0 | 1 | 0 | 0
  Calcium corrected for albumin - increased: baseline Grade 0 to maximum post-baseline Grade 1 | 0 | 9 | 0 | 0
  Creatinine - increased: baseline Grade 0 to maximum post-baseline Grade 1 | 3 | 5 | 1 | 2
  Creatinine - increased: baseline Grade 0 to maximum post-baseline Grade 2 | 1 | 2 | 0 | 0
  Creatinine - increased: baseline Grade 0 to maximum post-baseline Grade 3 | 0 | 0 | 0 | 1
  Creatinine - increased: baseline Grade 1 to maximum post-baseline Grade 2 | 0 | 1 | 0 | 0
  Glucose - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 0 | 3 | 0 | 2
  Lactate dehydrogenase - increased: baseline Grade 0 to maximum post-baseline Grade 1 | 3 | 22 | 3 | 4
  Lactate dehydrogenase - increased: baseline Grade 1 to maximum post-baseline Grade 0 | 1 | 0 | 0 | 0
  Potassium - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 3 | 4 | 2 | 1
  Potassium - decreased: baseline Grade 0 to maximum post-baseline Grade 3 | 0 | 0 | 0 | 1
  Potassium - decreased: baseline Grade 1 to maximum post-baseline Grade 0 | 0 | 1 | 1 | 0
  Potassium - increased: baseline Grade 0 to maximum post-baseline Grade 1 | 1 | 4 | 0 | 1
  Potassium - increased: baseline Grade 0 to maximum post-baseline Grade 2 | 0 | 4 | 1 | 1
  Sodium - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 7 | 10 | 3 | 3
  Sodium - decreased: baseline Grade 0 to maximum post-baseline Grade 2 | 1 | 2 | 0 | 1
  Sodium - decreased: baseline Grade 0 to maximum post-baseline Grade 3 | 0 | 1 | 0 | 0
  Sodium - decreased: baseline Grade 1 to maximum post-baseline Grade 0 | 0 | 1 | 1 | 0
  Sodium - decreased: baseline Grade 1 to maximum post-baseline Grade 2 | 0 | 1 | 0 | 0
  Total bilirubin - increased: baseline Grade 0 to maximum post-baseline Grade 1 | 1 | 2 | 0 | 0
  Total bilirubin - increased: baseline Grade 0 to maximum post-baseline Grade 3 | 1 | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Grade Shift From Baseline to Maximum Post-Baseline in Hematology Parameters Assessed by NCI CTCAE
Description: In this outcome measure, number of participants with baseline laboratory hematology values as per NCI-CTCAE grade (grade 0= within normal limits, grade 1=mild, grade 2=moderate, grade 3= severe, grade 4= life-threatening) and corresponding changes or shift to the worst CTC grades post baseline were presented. Laboratory parameters evaluated: hemoglobin- decreased and increased, leukocytes- decreased and increased, lymphocytes- decreased and increased, neutrophils decreased, platelets decreased. Baseline was defined as last non-missing grade before first dose of study treatment and worst post-baseline value defined as worst value post study treatment. Only those categories in which at least 1 participant had data in any reporting group were reported.
Time Frame: Baseline up to approximately 15.8 months
Population: The safety analysis set included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Number analyzed (Participants) | 21 | 39 | 9 | 8
Participants
  Hemoglobin - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 7 | 11 | 4 | 2
  Hemoglobin - decreased: baseline Grade 0 to maximum post-baseline Grade 2 | 0 | 0 | 2 | 1
  Hemoglobin - decreased: baseline Grade 0 to maximum post-baseline Grade 3 | 0 | 0 | 1 | 1
  Hemoglobin - decreased: baseline Grade 1 to maximum post-baseline Grade 2 | 3 | 1 | 0 | 3
  Hemoglobin - decreased: baseline Grade 1 to maximum post-baseline Grade 3 | 1 | 0 | 1 | 1
  Hemoglobin - decreased: baseline Grade 2 to maximum post-baseline Grade 1 | 0 | 1 | 0 | 0
  Hemoglobin - increased: baseline Grade 0 to maximum post-baseline Grade 1 | 0 | 2 | 0 | 0
  Leukocytes - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 1 | 3 | 2 | 4
  Leukocytes - decreased: baseline Grade 0 to maximum post-baseline Grade 2 | 0 | 0 | 1 | 0
  Leukocytes - decreased: baseline Grade 0 to maximum post-baseline Grade 3 | 0 | 0 | 1 | 0
  Lymphocytes - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 2 | 9 | 1 | 1
  Lymphocytes - decreased: baseline Grade 0 to maximum post-baseline Grade 2 | 4 | 0 | 2 | 0
  Lymphocytes - decreased: baseline Grade 0 to post-baseline Grade 3 | 1 | 1 | 1 | 0
  Lymphocytes - decreased: baseline Grade 0 to maximum post-baseline Grade 4 | 0 | 0 | 1 | 0
  Lymphocytes - decreased: baseline Grade 1 to maximum post-baseline Grade 2 | 1 | 1 | 0 | 1
  Lymphocytes - decreased: baseline Grade 1 to maximum post-baseline Grade 3 | 0 | 0 | 0 | 1
  Lymphocytes - decreased: baseline Grade 2 to maximum post-baseline Grade 3 | 0 | 2 | 1 | 0
  Lymphocytes - decreased: baseline Grade 3 to maximum post-baseline Grade 4 | 0 | 0 | 0 | 1
  Lymphocytes - increased: baseline Grade 0 to maximum post-baseline Grade 2 | 0 | 1 | 0 | 0
  Neutrophils - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 1 | 2 | 0 | 0
  Neutrophils - decreased: baseline Grade 0 to maximum post-baseline Grade 2 | 0 | 0 | 2 | 1
  Neutrophils - decreased: baseline Grade 0 to maximum post-baseline Grade 3 | 0 | 0 | 1 | 0
  Platelets - decreased: baseline Grade 0 to maximum post-baseline Grade 1 | 1 | 1 | 4 | 3

5. Secondary Outcome: Number of Participants With Treatment Interruptions, Dose Reductions, Treatment Discontinuations Due to Adverse Events
Description: An AE is defined as any untoward medical occurrence in participant/clinical investigational participant administered medicinal product which doesn't necessarily have causal relationship with treatment. Number of participants with dose interruption (SEA-CD40 treatment being temporarily stopped), dose reduction (SEA-CD40 decrease in dose) and dose discontinuation (SEA-CD40 treatment permanently stopped) due to adverse events were reported in this outcome measure.
Time Frame: From first dose of the study treatment (Day 1) up to approximately 18.5 months
Population: The safety analysis set included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Number analyzed (Participants) | 21 | 39 | 9 | 8
Participants
  Treatment interruptions | 1 | 5 | 2 | 1
  Dose reductions | 0 | 0 | 0 | 0
  Treatment discontinuations | 2 | 0 | 2 | 1

6. Secondary Outcome: Disease Control Rate (DCR) Per Investigator Assessment
Description: DCR is defined as the percentage of participants who achieved a confirmed CR or PR according to RECIST v1.1 as assessed by the investigator or met the stable disease (SD) criteria at least once after start of study treatment at a minimum interval of 5 weeks. CR: disappearance of all target, non-target lesions, all lymph nodes must be non-pathological in size (<10 mm short axis), PR: at least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters persistence of one or more non-target lesions. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase in lesions to qualify for progressive disease (PD) referring smallest sum diameter, PD: at least 20% increase (including absolute increase of at least 5 mm) in sum of diameters of target lesions, taking reference smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From the first dose of study treatment until the first documented CR, PR or SD or new anticancer therapies or death, whichever occurred first (maximum up to 15.2 months)
Population: The RE analysis set included all participants with measurable disease at baseline who received any amount of study drug and had at least one post-baseline disease assessment per RECIST v1.1 or discontinued study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Number analyzed (Participants) | 21 | 39 | 9 | 8
Percentage of participants | 48 [25.7 to 70.2] | 62 [44.6 to 76.6] | 67 [29.9 to 92.5] | 88 [47.3 to 99.7]

7. Secondary Outcome: Duration of Response (DOR) Per Investigator Assessment
Description: DOR: time from first documentation of OR (confirmed CR or PR) to first documentation of PD or death due to any cause, whichever occurred first. Per RECIST v1.1- CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: >=30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. Participants with no PD and were still on study at time of analysis or were removed from study prior to documentation of PD were censored at last disease assessment documenting absence of PD. Participants who started new anticancer treatment prior to documentation of PD were censored at last disease assessment prior to start of new treatment. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must demonstrate absolute increase of 0.5 cm. Appearance of 1 or more new lesions. Kaplan-Meier method was used.
Time Frame: From the first documentation of CR or PR to PD or death due to any cause or censoring, whichever occurred first (maximum up to 11.1 months)
Population: The RE analysis set included all participants with measurable disease at baseline who received any amount of study drug and had at least one post-baseline disease assessment per RECIST v1.1 or discontinued study treatment. Here, ''Overall Number of Participants Analyzed'' signifies participants with confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Number analyzed (Participants) | 0 | 2 | 4 | 2
Months |  | NA [5.6 to NA] — Median and upper limit of the 95% confidence interval was not estimable due to insufficient number of participants with events. | 11.1 [9.9 to NA] — Upper limit of the 95% confidence interval was not estimable due to insufficient number of participants with events. | 2.1 [NA to NA] — Lower and upper limit of the 95% confidence interval was not estimable due to insufficient number of participants with events.

8. Secondary Outcome: Progression Free Survival (PFS) Per Investigator Assessment
Description: PFS is defined as time from start of study treatment to first documentation of PD by RECIST v1.1 or death due to any cause, whichever occurred first. Participants with no PD and were still on study at time of analysis or who were removed from study prior to documentation of PD were censored at the date of last disease assessment documenting absence of PD. Participants who started new anticancer treatment prior to documentation of PD were censored at date of last disease assessment prior to start of new treatment. PD: At least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study (this included baseline sum if that is the smallest on study). In addition to relative increase of 20%, the sum must also demonstrate an absolute increase of at least 0.5 cm. Appearance of one or more new lesions was also considered progression. Kaplan-Meier method was used.
Time Frame: From first dose of study treatment to the date of PD or death due to any cause or censoring, whichever occurred first (maximum up to 13.9 months)
Population: The full analysis set (FAS) includes all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Number analyzed (Participants) | 21 | 39 | 9 | 8
Months | 1.6 [1.4 to 2.9] | 4.0 [1.4 to 8.2] | 13.8 [1.4 to NA] — Upper limit of the 95% confidence interval was not estimable due to insufficient number of participants with events. | 5.5 [1.4 to NA] — Upper limit of the 95% confidence interval was not estimable due to insufficient number of participants with events.

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the start of study treatment to date of death due to any cause. In the absence of death, survival time was censored at the last date the participant was known to be alive. Kaplan-Meier method was used for analysis.
Time Frame: From start of study treatment to death due to any cause or censoring date (maximum up to 23.6 months)
Population: The FAS includes all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
Number analyzed (Participants) | 21 | 39 | 9 | 8
Months | 11.0 [5.3 to 18.7] | NA [16.7 to NA] — Median and upper limit of the 95% confidence interval was not estimable due to insufficient number of participants with events. | 18.0 [2.5 to NA] — Upper limit of the 95% confidence interval was not estimable due to insufficient number of participants with events. | NA [3.2 to NA] — Median and upper limit of the 95% confidence interval was not estimable due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: From first dose of the study treatment (Day 1) up to approximately 18.5 months for SAEs, 16.5 months for non-SAEs and 23.6 months for death
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. Event may be categorised as serious in 1 participant and non-serious in other, or participant may have experienced both serious and non-serious event. The safety analysis set included all participants who received any amount of study drug.
Arm/Group | Cohort 1: Relapsed/Refractory Melanoma | Cohort 2: Uveal Melanoma | Cohort 4: NSCLC, PD-L1 1-49% | Cohort 5: NSCLC, PD-L1 < 1%
All-Cause Mortality (participants affected / at risk) | 11/21 | 8/39 | 3/9 | 1/8
Serious Adverse Events (participants affected / at risk) | 4/21 | 5/39 | 5/9 | 5/8
Other Adverse Events (participants affected / at risk) | 17/21 | 37/39 | 8/9 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Relapsed/Refractory Melanoma (N=21) | Cohort 2: Uveal Melanoma (N=39) | Cohort 4: NSCLC, PD-L1 1-49% (N=9) | Cohort 5: NSCLC, PD-L1 < 1% (N=8)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Relapsed/Refractory Melanoma (N=21) | Cohort 2: Uveal Melanoma (N=39) | Cohort 4: NSCLC, PD-L1 1-49% (N=9) | Cohort 5: NSCLC, PD-L1 < 1% (N=8)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 4 (6) | 6 (9)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 6 (6) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 8 (10) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 15 (16) | 1 (2) | 3 (3)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 9 (10) | 3 (5) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (15) | 16 (28) | 7 (9) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Vomiting (Gastrointestinal disorders) | 6 (8) | 3 (4) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 6 (8) | 11 (16) | 2 (4) | 3 (4)
Fatigue (General disorders) | 4 (5) | 24 (32) | 7 (9) | 3 (4)
Malaise (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (5) | 2 (3) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 12 (17) | 11 (23) | 3 (6) | 4 (5)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 6 (8) | 1 (6) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (5) | 1 (4) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 7 (7) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (4) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (4) | 2 (2) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (4) | 3 (4) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3) | 0 (0) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (5) | 6 (6) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (10) | 1 (1) | 1 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 5 (5) | 3 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 13 (18) | 4 (4) | 2 (3)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Vulvovaginal rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (9) | 1 (1) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 1 (1) | 3 (3)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 4 (4) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 5 (6) | 3 (3) | 2 (2) | 2 (3)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT04993677/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT04993677/SAP_001.pdf